CLINICAL TRIAL: NCT01975584
Title: Neuroendocrine and Immune Response to Stress in Schizophrenia
Acronym: TSST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Deanna Kelly, Pharm.D., BCPP, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-00055151
Record Dates: First submitted 2013-10-18; First posted 2013-11-04 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trier Social Stress Test (Experimental): Participants will participate in a standardized role play (Trier Social Stress Test ). A role play is pretending to be in a certain situation. A research staff member will describe the role play, during which teh participant will act out a scene. Participants will be asked to imagine that they are in a certain role with several other research team members who will also participate in the role play. Participants will also be asked to do some math problems without using paper or pencil.
  Interventions: Behavioral: Trier Social Stress Test

INTERVENTIONS:
Behavioral: Trier Social Stress Test — Participants will participate in a standardized role play (Trier Social Stress Test ). A role play is pretending to be in a certain situation. A research staff member will describe the role play, during which teh participant will act out a scene. Participants will be asked to imagine that they are in a certain role with several other research team members who will also participate in the role play. Participants will also be asked to do some math problems without using paper or pencil.

SUMMARY:
This is a pilot study. We are testing the physiologic, immune and chemical responses to stress. We believe the results of all measures to stress will be blunted in schizophrenia compared to healthy controls. We will test sex, early life stress and other factors on the relationship to a stress response.

DETAILED DESCRIPTION:
The proposed study examines the response of neuroimmune and inflammatory responses to a stress in both men and women with a DSM-IV diagnosis of schizophrenia or schizoaffective disorder. The measurements include stress hormones or other elements in the blood which indicate stress . Early childhood trauma/stress (ELS) information will be collected so we can examine differences in those with trauma histories vs. those with none by sex. There will be one visit for screening before the testing visit. The sample will consist of up to 45 clinically stable inpatients and outpatients with DSM-IV schizophrenia or schizoaffective disorder, of which approximately 15 will be women. We will also enroll up to 45 healthy controls without a DSM-IV Axis I or II disorder. Prior to the study all subjects must meet inclusion and exclusion criteria including a medical history.

The (TSST) is a standard and widely used research assessment procedure that is used to reliably induce stress in human research participants. The TSST uses situations where people think they are being socially evaluated during an interview for a job. Participants are told they are competing with other people for this job, and their task is to convince interviewers that they are the best person for the job. Participants are told they have to prepare a speech, and complete a math challenge in their head.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder (schizophrenia group)
* No DSM-IV Axis I or II disorder (healthy control group)
* Caucasian or Non-Caucasian

Exclusion Criteria:

* History of Cushing's syndrome, adrenal deficiency, or any condition that may affect cortisol levels in the body.
* Use of steroids
* Pregnancy or lactation. Pregnancy will be determined by urine pregnancy test. Lactation will be determined through patient report.
* Untreated hypertension, cardiac arrthymias or medical condition that could not handle stress.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Aim 1) To examine neuroendocrine and physiologic response following a psychosocial stressor in people with schizophrenia and healthy controls. | 1 week
  We will administer the Trier Social Stress Test (TSST) and measure neuroendocrine values (plasma and salivary cortisol and adrenocorticotropic hormone (ACTH) and physiologic variables (heart rate, blood pressure) before during and after the TSST.

SECONDARY OUTCOMES:
To investigate neuroimmune and kynurenic acid modulation to a psychosocial stressor in people with schizophrenia and healthy controls | 1 week
  We will measure peripheral cytokine response (IL-6, IL1-Beta, TNF alpha) and kynruenic acid, kynurenine and pathway metabolites before, during and after the TSST.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, PharmD, BCPP, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu